CLINICAL TRIAL: NCT06869590
Title: Identification of Anti-HIF 1alpha Autoantibodies in Patients With Anorexia Nervosa and Characterization of Their Pathogenic Potential in Undernutrition-associated Hepatic Cytolysis
Acronym: HIAM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RCAPHM24_0497; 2025-A00018-41 (Other: IDRCB)
Record Dates: First submitted 2025-02-26; First posted 2025-03-11 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Hepatic Cytolysis
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patient with anorexia nervosa and anti-HIF1a autoantibody positivity (Experimental): When blood is drawn as part of the treatment, three additional dry tubes will be taken for the immunology laboratory (see study diagram). These three dry tubes will be used to test for 1/ anti-nuclear autoantibodies and those associated with hepatic autoimmune pathologies 2/ AAHIF and assess their pathogenic potential using techniques already developed. In the event of AAHIF positivity, a second sample will be taken between 12 and 16 weeks later to verify the persistence of autoantibodies: Visit 2. The third dry tube will be sent to the Biogénopole Biological Resource Center (CHU Timone, APHM).
  Interventions: Other: blood sampling; Other: blood sampling after 3-4 months
- Patient with anorexia nervosa and no anti-HIF1a autoantibody positivity (Experimental): When blood is drawn as part of the treatment, three additional dry tubes will be taken for the immunology laboratory (see study diagram). These three dry tubes will be used to test for 1/ anti-nuclear autoantibodies and those associated with hepatic autoimmune pathologies 2/ AAHIF and assess their pathogenic potential using techniques already developed. The third dry tube will be sent to the Biogénopole Biological Resource Center (CHU Timone, APHM).
  Interventions: Other: blood sampling
- Patient without anorexia nervosa and anti-HIF1a autoantibody positivity (Active Comparator): When blood is drawn as part of the treatment, three additional dry tubes will be taken for the immunology laboratory (see study diagram). These three dry tubes will be used to test for 1/ anti-nuclear autoantibodies and those associated with hepatic autoimmune pathologies 2/ AAHIF and assess their pathogenic potential using techniques already developed. In the event of AAHIF positivity, a second sample will be taken between 12 and 16 weeks later to verify the persistence of autoantibodies: Visit 2. The third dry tube will be sent to the Biogénopole Biological Resource Center (CHU Timone, APHM).
  Interventions: Other: blood sampling; Other: blood sampling after 3-4 months
- Patient without anorexia nervosa and no anti-HIF1a autoantibody positivity (Active Comparator): When blood is drawn as part of the treatment, three additional dry tubes will be taken for the immunology laboratory (see study diagram). These three dry tubes will be used to test for 1/ anti-nuclear autoantibodies and those associated with hepatic autoimmune pathologies 2/ AAHIF and assess their pathogenic potential using techniques already developed. The third dry tube will be sent to the Biogénopole Biological Resource Center (CHU Timone, APHM).
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — When blood is drawn as part of the treatment, three additional dry tubes will be taken for the immunology laboratory (see study diagram). These three dry tubes will be used to test for 1/ anti-nuclear autoantibodies and those associated with hepatic autoimmune pathologies 2/ AAHIF and assess their pathogenic potential using techniques already developed. The third dry tube will be sent to the Biogénopole Biological Resource Center (CHU Timone, APHM).
Other: blood sampling after 3-4 months — In the event of AAHIF positivity, a second sample will be taken between 12 and 16 weeks later to verify the persistence of autoantibodies: Visit 2.
  Arms: Patient with anorexia nervosa and anti-HIF1a autoantibody positivity; Patient without anorexia nervosa and anti-HIF1a autoantibody positivity

SUMMARY:
Anorexia nervosa (AN) is a psychiatric disorder belonging to the eating disorders (EDs). It is internationally recognized as a priority for improving health care. Among the markers of severity of undernutrition is hepatic cytolysis. Around 30-50% of patients with AN present with hepatic cytolysis, of variable intensity, and usually associated with severe undernutrition. In a previous study, we demonstrated the presence of autoantibodies against HIF1alpha (Hypoxic inducible Factor 1 alpha) in 22% of cases in a sample of patients with AN. HIF1alpha (HIF1a) is a major transcription factor involved in the regulation of satiety and hunger. These autoantibodies were positive in 80% of AN patients with hepatic cytolysis. Taken together, these data led us to hypothesize an anti-HIF1a autoimmune mechanism in AN, potentially involved in the patients' hepatic cytolysis.

This pioneering study, demonstrating the existence of anti-HIF1a autoantibodies, was carried out on a population of 18 patients with AN. To extend investigator's hypothesis, these results need to be confirmed on a larger number of patients, thus increasing the number of patients with AN and hepatic cytolysis. To determine the relevance of these autoantibodies in AN, "healthy" subjects and patients without AN but with hepatic cytolysis should be tested in parallel. Finally, the in vitro pathogenic potential of autoantibodies can be confirmed on a larger scale and studied in greater detail.

The main aim of our study is to evaluate the association between the presence of anti-HIF1a autoantibodies (AAHIF) and that of hepatic cytolysis in patients with anorexia nervosa and undernutrition.

This study is a prospective, cross-sectional, descriptive, multicenter, 2-arm study.

250 patients will be included. Experimental group (n=100)

* Patients with anorexia nervosa and undernutrition with hepatic cytolysis (CH) (n=70)
* Patients with anorexia nervosa and undernutrition without hepatic cytolysis (n=30) Comparator control groups (n=150)
* Control patients under 18 years of age, treated at the CHU de la Timone for scheduled non-inflammatory surgery (orthopedic, ENT, etc.) (n=50): Minor patients
* Patients (children and adults) with hepatic cytolysis without anorexia nervosa (n=50): Patients without AN with CH
* Samples from French blood donation establishment: control group consisting of biological blood samples from healthy individuals from the Etablissement Français du Sang (n=50)

ELIGIBILITY:
Inclusion Criteria:

Experimental group:

* Male or female, 6 to 65 years of age
* Anorexia nervosa diagnosed according to DSM-5 criteria
* Presence of undernutrition according to HAS 2019 criteria
* Patient having received information about the study and having signed an informed consent form
* Beneficiary or beneficiary of a social security scheme

Control group:

* Minor patients :

  * Male or female strictly under 18 years of age
  * Patients undergoing scheduled non-inflammatory surgery (orthopedic, ENT, etc.)
  * Patients who have been informed about the study and have signed an informed consent form.
  * Patients who are beneficiaries or entitled beneficiaries of a social security scheme.
* Patients without anorexia with livers cytolysis :

  * Male or female between 18 and 65 years of age
  * With hepatic cytolysis determined by an ALT value at least equal to twice the normal value
  * Patient having received information about the study and having signed an informed consent form
  * Patient who is a beneficiary or eligible beneficiary of a social security scheme.
* samples Etablissement Français de don de sang: no specific criteria

Exclusion Criteria:

* Patient in a period of exclusion from another research protocol at the time consent is signed.
* Opposition of patient and parents or legal guardians
* Psychiatric disorder preventing patient consent to study
* Person unable to understand the French language
* Subjects covered by articles L1121-5 to 1121-8 of the French Public Health Code (minors, adults under guardianship or trusteeship, patients deprived of their liberty, pregnant or breast-feeding women).

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-11-24 (Estimated); Primary Completion 2027-05-24 (Estimated); Study Completion 2029-05-24 (Estimated)

PRIMARY OUTCOMES:
Determination of anti-HIF1a autoantibodies (AAHIF) in comparison with the presence of hepatic cytolysis in patients with anorexia nervosa and undernutrition | From enrollment to the end of study at 36 months
  Comparison of the prevalence of anti-HIF1a autoantibodies (AAHIF) in patients with AM according to the presence or absence of hepatic cytolysis.

SECONDARY OUTCOMES:
Rate of AAHIF in a population of healthy subjects | From enrollment to the end of the study at 36 months
Rate of AAHIF in patients without anorexia nervosa and with hepatic cytolysis. | From enrollment to the end of the study at 36 months
Rate of AAHIF in patients with anorexia nervosa and suffering from malnutrition | From enrollment to the end of the study at 36 months
Rate of AAHIF according to clinico-biological criteria for AOS identified in routine care | From enrollment to the end of the study at 36 months
  age, sex, type of AN (pure or mixed restrictive, restrictive and hyperphagic/purgative), duration of disorders, attitudes and behaviors related to AN (assessed by the Eating Disorder Inventory 2 EDI 2 questionnaire), weight, BMI, weight loss in 1 month, weight loss in 6 months or since onset of illness, severity of undernutrition, presence of problematic physical hyperactivity (assessed by the Exercise Dependence Scale-Revised EDSR questionnaire), presence of amenorrhea, use of enteral nutrition, associated treatments, leukocytes, neutrophils, lymphocytes, hemoglobin, platelets, creatinine, urea, AST, ALT, GGT, fasting blood glucose, PT, albumin, pre-albumin (transthyretin), vitamin B12, folate, vitamin D, ferritin.
Pathogenic potential in vitro of AAHIF in hepatic cytolysis | From enrollment to the end of the study at 36 months
  Functional effects of the purified AAHIF fraction on hepatocyte cell lysis and its impact on HIF1a-dependent signaling.

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux De Marseille, Marseille, France